CLINICAL TRIAL: NCT02765217
Title: Effect of Lactobacillus Reuteri DSM 17938 to Prevent Antibiotic-associated Diarrhea in Children: Prospective, Multi-center, Randomize, Parallel Group Placebo Controlled Clinical Trial
Brief Title: Effect of Lactobacillus Reuteri DSM 17938 to Prevent Antibiotic-associated Diarrhea in Children
Acronym: PEARL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Hacettepe University (Other); Acıbadem University School of Medicine (Other); Umraniye Education and Research Hospital (Other Government); Sisli Hamidiye Etfal Training and Research Hospital (Other); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Ege University Medical School (Other); Yuzuncu Yil University (Other); Goztepe Training and Research Hospital (Other); Erzurum Regional Training & Research Hospital (Other Government); Namik Kemal University (Other)
Responsible Party: Principal Investigator, Ener Cagri DINLEYICI, Professor in Pediatrics, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROBAGE006
Record Dates: First submitted 2016-05-02; First posted 2016-05-06 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Antibiotic Associated Diarrhea
Keywords: Antibiotic associated diarrhea; Children; Prevention; Lactobacillus reuteri DSM 17938; Probiotic
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study group 1 (Experimental): Amoxicilline-clavulanic acid (50-90 mg/kg/day, twice daily) and Lactobacillus reuteri DSM 17938 (5 drops per day, same time with the first dose of antibiotics).
  Study Group 1a will received L. reuteri for 10-14 days. Study Group 1b will received L. reuteri for 21 days.
  Interventions: Drug: Lactobacillus reuteri DSM 17938; Drug: Amoxicillin-Clavulanic Acid
- Study group 2 (Placebo Comparator): Amoxicillin-clavulanic acid (50-90 mg / kg / day) and placebo ( 5 drops per day, same time with the antibiotics) Study Group 2a will received placebo for 10-14 days. Study Group 2b will received placebo for 21 days.
  Interventions: Drug: Placebo; Drug: Amoxicillin-Clavulanic Acid
- Study group 3 (Experimental): Amoxicilline-clavulanic acid (50-90 mg/kg/day, twice daily) and Lactobacillus reuteri DSM 17938 (2 x 5 drops per day) Study Group 3a will received L. reuteri for 10-14 days. Study Group 3b will received L. reuteri for 21 days.
  Interventions: Drug: Lactobacillus reuteri DSM 17938; Drug: Amoxicillin-Clavulanic Acid
- Study group 4 (Placebo Comparator): Amoxicillin-clavulanic acid (50-90 mg / kg / day) and placebo ( 2 x 5 drops per day, same time with the antibiotics) Study Group 4a will received placebo for 10-14 days. Study Group 4b will received placebo for 21 days.
  Interventions: Drug: Placebo; Drug: Amoxicillin-Clavulanic Acid

INTERVENTIONS:
Drug: Lactobacillus reuteri DSM 17938 — Comparison the effects of Lactobacillus reuteri DSM 17938 and placebo for prevention of antibiotic associated diarrhea and also plan to compare the duration of treatment for on efficacy.
  Other Names: BioGaia
  Arms: Study group 1; Study group 3
Drug: Placebo — Comparison the effects of Lactobacillus reuteri DSM 17938 and placebo for prevention of antibiotic associated diarrhea and also plan to compare the duration of treatment for on
  Arms: Study group 2; Study group 4
Drug: Amoxicillin-Clavulanic Acid — All study patients will received amoxicillin-clavulanic acid at the dose of 50-90 mg/kg/day.
  Other Names: Co-amoxilav

SUMMARY:
Recent studies showed that intestinal microbiota consist more than thousand bacteria, and these microorganisms play the role as balance and continuity of the anatomical and functional integrity gastrointestinal tract. Chronic diseases, nutritional factors, lifestyle factors and medications including antibiotics changes the host microbiota in short or long-term period. Antibiotics are the most commonly used drugs in pediatrics routine practice. Although frequency and severity of side effects alter the choice of drug, mild complications may be taken into consideration for treatment by a physician in the profit and loss balance. Our study group (PROBAGE Working Group) have been recently showed that Lactobacillus reuteri DSM 17938 reduced the duration of diarrhea in children with acute infectious diarrhea, and are safe and well-tolerated. In this study the investigators aim to evaluate the potential effect of Lactobacillus reuteri DSM 17938 on the prevention of antibiotic associated diarrhea in children.

DETAILED DESCRIPTION:
Recent studies showed that intestinal microbiota consist more than thousand bacteria, and these microorganisms play the role as balance and continuity of the anatomical and functional integrity gastrointestinal tract. Chronic diseases, nutritional factors, lifestyle factors and medications including antibiotics changes the host microbiota in short or long-term period. Antibiotics are the most commonly used drugs in pediatrics routine practice. Although frequency and severity of side effects alter the choice of drug, mild complications may be taken into consideration for treatment by a physician in the profit and loss balance.

Antibiotic-associated diarrhea is one of the side effects that occur during antibiotic use, the frequency varies according to region and antibiotic type. Aminopenicillins, cephalosporins and clindamycin antibiotics has been identified as the most affected group of antibiotic-associated diarrhea. Development of antibiotic associated diarrhea are associated with the intestinal microbiota balance , the mucosal integrity and changes of vitamin / mineral metabolism 3. Majority cases with antibiotic associated diarrhea admit with the complaints of abdominal crampy pain and diarrhea while pseudomembranous enterocolitis, in severe cases, even death have been reported. Antibiotic-associated diarrhea can be occur during antibiotic treatment but may seen at 2-3 weeks later after termination of treatment. Broad-spectrum antimicrobial agents have been related 11-40% of antibiotic associated diarrhea cases in children.

In Turkey there are no large studies on the frequency of antibiotic associated diarrhea in children, but antibiotics are the most commonly used drug classes in childhood. The use of broad-spectrum antibiotics, which creates more risk than narrow-spectrum antibiotics, and the highest risk have been observed during use of clindamycin, cephalosporins and fluoroquinolones. However, there is no consensus about which antibiotics which are high risk or which have significant negative impact on the microbiota. Antibiotic-associated diarrhea, has been shown to increase the growth of enteropathogens after antibiotic use.

In particular, Clostridium difficile (C. difficile) infections are the most common infections which related with antibiotic associated diarrhea 2. Although C. difficile diarrhea mostly occurs in adults and hospitalized immunocompromised patients, it can be seen in children.

C. difficile leads to mild diarrhea to pseudomembranous colitis according to toxins. C. difficile associated 10-20% of all antibiotic-associated diarrhea forms and can be seen until after eight weeks of treatment with antibiotics. Antibiotics disrupt the integrity of the normal colonic mucosa, affect carbohydrate metabolism as a result of antimicrobial activity in the colon leads to the development of osmotic diarrhea and pathogenic bacteria associated diarrhea. The slowing of the metabolism of carbohydrates results in the reduction of short-chain fatty acids in the intestinal lumen and cause accumulation of carbohydrates which can not be absorbed. Besides the harm normal microbiota have provided the protective barrier and intestinal system becomes sensitive to resistant microorganisms. Reduction of intestinal lumen and in the number of Bacteroides and Bifidobacteria strains of facultative anaerobes (Fusobacterium the Clostridia, Eubacteria) results in the increase. Antibiotic-associated diarrhea, alongside a negative effect on the quality of life of the host, the cost of treatment in patients hospitalized in the hospital and also negatively affects the length of stay.

In case of outpatient treatment, or in hospitalized patients, antibiotic treatment usually is terminated or is changed, it affects the success of the treatment in this case and leads to a longer stay in hospital. Especially the long-term hospitalization in the intensive care unit at the hospital caused by an increase in the risk of nosocomial infections and has been shown to cause mortality 14.

In case of diarrhea in patients treated ambulatory during treatment if the patient's symptoms also declined, antibiotic treatment is interrupted by family. If cases can result in use therefore again brought to the physician if the physician broader spectrum antibiotics or parenteral drugs.

In studies with probiotics, some of the probiotic strains of antibiotic-associated diarrhea development when used in combination with antibiotics it has been shown to be significantly reduced. Harvard / Yale probiotic Workshop Group, World Gastroenterology Organization in the prevention of antibiotic associated diarrhea probiotic strains showed that the level of evidence A1. However, probiotics effects are strain specific. Although Saccharomyces boulardii and Lactobacillus GG are well known strains for prevention of antibiotic associated diarrhea, knowledge about the Lactobacillus reuteri DSM 17938 is limited.

Our study group (PROBAGE Working Group) have been recently showed that Lactobacillus reuteri DSM 17938 reduced the duration of diarrhea in children with acute infectious diarrhea, and are safe and well-tolerated. In this study the investigators aim to evaluate the potential effect of Lactobacillus reuteri DSM 17938 on the prevention of antibiotic associated diarrhea in children.

ELIGIBILITY:
Inclusion Criteria:

• Children receiving amoxicilline-clavulanic acid (50-90 mg/kg/day, twice daily) due to acute otitis media or acute sinusitis

Exclusion Criteria:

* Receiving antibiotic and/or probiotic, 8 weeks before the study
* Chronic gastrointestinal system disorders
* Congenital anomalies
* Chronic diseases
* Chemotherapy and radiotherapy
* Pregnancy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1325 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic associated diarrhea | 8 weeks time period after 1st day of antibiotic use
  The frequency and consistency of the stools were recorded daily according to Bristol score; a score <5 is described as normalization of stool and score equal or above 5 defined as diarrhea. Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug, Graded According to NCI CTCAE Version 3.0

SECONDARY OUTCOMES:
Incidence of antibiotic associated diarrhea during antibiotic treatment | 10-14 days (depends on the antibiotic treatment)
  The frequency and consistency of the stools were recorded daily according to Bristol score; a score <5 is described as normalization of stool and score equal or above 5 defined as diarrhea.
Incidence of antibiotic associated diarrhea after antibiotic treatment | From 11-15th days of intervention to 56 days
  The frequency and consistency of the stools were recorded daily according to Bristol score; a score <5 is described as normalization of stool and score equal or above 5 defined as diarrhea.
Evaluation of antibiotic-associated diarrhea in patients who developed diarrhea severity | 56 days
  Presence of dehydration, requiring medical care, requiring hospitalization, Vesikari scale score
The frequency of other gastrointestinal symptoms other than diarrhea during the study (will be evaluated using the Gastrointestinal Symptom Rating Score) | 56 days
  The Gastrointestinal Symptoms Rating Score, is a disease-specific instrument of 15 items combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. The Gastrointestinal Symptom Rating Score has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Etfal Training and Research Hospital,, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Dinleyici EC, Ozen M, Guven S, Dalgic N, Karbuz A, Sutcu M, Turel O, Oz FN, Kirli U, Yasar Durmus S, Yazar AS, Cakin ZE, Vandenplas Y, Kara A. Effect of Limosilactobacillus reuteri DSM17938 to prevent antibiotic-associated diarrhea in children: prospective, multi-center, randomized, placebo-controlled clinical trial (PEARL Study). Eur J Pediatr. 2025 Jun 9;184(7):408. doi: 10.1007/s00431-025-06249-8. PMID 40488914